CLINICAL TRIAL: NCT03522753
Title: Staple Versus Suture Closure for Foot and Ankle Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Resolving database issues
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ashish Shah, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB-300001258
Record Dates: First submitted 2018-05-01; First posted 2018-05-11 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Incision; Foot Ankle Injuries
MeSH Terms: conditions — Surgical Wound | interventions — Sutures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The resident/fellow performing closure will know what has been done for their patient, but blinded to other participants. Splints or other dressings will cover the closure. Patients will be physically "blinded" (i.e. eye cover) during the removal procedure. Patients and observers will assess scar appearance. "Observers" are the blinded surgeon or other blinded medical personnel (nurse, research assistant, CRNP, or resident/fellow who was not involved).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Staples (Experimental): For short single incisions, these patients will receive superficial closure using only metal skin staples. Closure will be performed by resident or fellow involved in the case.
  Interventions: Device: Metal skin staples
- Suture (Active Comparator): For short single incisions, these patients will receive superficial closure using only nylon sutures. No metal skin staples will be used. Closure will be performed by resident or fellow involved in the case.
  Interventions: Device: Nylon sutures
- Half Staple Half Suture (Other): Some patients will receive both nylon sutures and metal skin staples for superficial closure. If multiple incisions are involved, each incision will count as 1 in the alternation method (i.e. toe 1 will be all sutures, then toe 2 will be all staples). For long incisions, closure will alternate between nylon sutures and metal skin staples on the part of the incision which is closer (more proximal) or farther away (more distal) from the rest of the body.
  Interventions: Device: Metal skin staples; Device: Nylon sutures

INTERVENTIONS:
Device: Metal skin staples — Routine closure methods/material for surgical wounds
  Other Names: metal clips; skin clips; staples
  Arms: Half Staple Half Suture; Staples
Device: Nylon sutures — Routine closure methods/material for surgical wounds
  Other Names: sutures
  Arms: Half Staple Half Suture; Suture

SUMMARY:
This study aims to determine if staples or sutures are better for the closure of uncomplicated foot and ankle surgeries. Currently, most surgeons base their choice for closure on previous teaching from a mentor during fellowship or personal experience. There is no standard of care for closure material on hand surgeries to date. This study will prospectively randomize patients to have either staple or suture wound closure if they have a short incision. In surgeries with longer incisions (i.e. 5+ cm), or multiple incisions on similar sites (i.e. bilateral operations, multiple toes), patients will have half sutures and half staple closure. The three primary measured outcomes will be: pain upon suture/staple removal, time to place and remove sutures vs. staples, and scar formation.

DETAILED DESCRIPTION:
The material used for closure of surgical incision is often considered "dealer's choice" and usually is chosen from one (or a combination) of the following techniques: subcutaneous absorbable sutures, interrupted simple/mattress dermal sutures, or dermal staples. Factors that are typically taken into consideration include anatomic location, amount of tension involved in closure, shape of the incision and integrity of the skin involved in the closure, need for cosmesis, and surgeon comfort/past experience with different closure techniques.

Previous randomized controlled trials, as well as meta-analyses, have analyzed sutures versus staples in orthopaedic surgeries, but often exclude foot and ankle surgeries as incisions are typically small and require more delicate closures. In RCTs involving other areas of the body, staples have been found to result in less wound infection and less time to insert/remove compared to sutures. They were also comparable to sutures in cosmetic result and patient satisfaction. These results are not known for surgeries of the foot and ankle.

Both sutures and staples are routinely used during a typical foot and ankle surgery, without significant risk of wound dehiscence or complications.

This study aims to determine if staples or sutures are better for the closure of uncomplicated foot and ankle surgeries. Currently, most surgeons base their choice for closure on previous teaching from a mentor during fellowship or personal experience. There is no standard of care for closure material on hand surgeries to date. This study will prospectively randomize patients to have either staple or suture wound closure if they have a short incision. In surgeries with longer incisions (i.e. 5+ cm), or multiple incisions on similar sites (i.e. bilateral operations, multiple toes), patients will have half sutures and half staple closure. The three primary measured outcomes will be: pain upon suture/staple removal, time to place and remove sutures vs. staples, and scar formation.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Scheduled to undergo any elective foot or ankle procedures with one of our included surgeons investigators during the approved protocol period.
* Patients with comorbidities such as rheumatoid arthritis, diabetes, and other systemic diseases will still be included so long as they are not considered uncontrolled or immunocompromised.
* In patients with rheumatoid arthritis, the usual protocol for discontinuing disease-modifying antirheumatic drugs (DMARDs) prior to surgery will be continued as done per each surgeon's protocol.
* Patients undergoing urgent surgery (e.g. within a few days of the inciting event, such as a traumatic fracture) will be considered for the study.

Exclusion Criteria:

* Patients under 18 years old
* Patients who are not competent to give consent for themselves, or to read and answer questions about their scar formation (proxies will not be allowed);
* Any surgery that requires a non-linear surgical incision;
* Previous surgery(ies) on the same area;
* Known history of keloid/abnormal scar formation;
* Patients with uncontrolled diabetes (as documented by ICD-9 codes 250.x2 or 250.x3);
* Patients who are immunocompromised (i.e. HIV/AIDS+ patients, patients who have had a previous organ transplantation, patients who have been diagnosed with an immunodeficiency syndrome- congenital or acquired, as a result of immunomodulatory medication secondary to autoimmune disease, or undergoing current chemotherapy for cancer).
* Patients undergoing emergent surgery will not be considered for the study.
* Patients who have had a previous allergic or adverse reaction to any of the suture/staple materials we plan to use will not be included.
* If the closure requires multiple layers of sutures (i.e. subcutaneous layers, deep dermal layers) in addition to the usual closing staples/sutures which are through the skin, the patient will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Pain on removal | At time of device removal (10-14 days post-op)
  Visual Analog Scale (VAS) Pain Score; Scale 0-10, where 0=no pain and 10=worst possible pain

SECONDARY OUTCOMES:
Time to place and remove | At time of surgery and at time of device removal (10-14 days post-op)
  Time in seconds to place and remove device
Scar formation | At time of device removal (10-14 days post-op), at 6 weeks, 3 months, and 1 year post-op
  Modified Patient and Observer Scar Assessment Scale (POSAS) Questionnaire. This questionnaire rates scar formation using two total scores, each between 6-60 points (lower score is better), one completed by the patient (patient scale) and one by an observer (observer scale). The total score for each scale is the sum of 6 equally weighted questionnaire items (each scoring 1-10 points; lower score is better). In addition, both patient and observer give overall opinion of scarring, on a 1-10 scale; lower score is better. Overall opinions reported separately from total scores.

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Shah, MD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No
Only investigators involved in the research protocol will have knowledge of any patient involvement. Research meetings will be closed to any other participants and will be conducted in a closed office setting away from passersby. Documents with any kind of patient information/involvement will be kept on a secure, password protected server that cannot be accessed by those not involved with the protocol. Similarly, consent forms will be kept in the office of the principal investigator in a locked drawer. Research data will be stored on a secure server which is only accessible by investigators who have been individually allowed access to the project. Only aggregate or unidentifiable data will be published.